CLINICAL TRIAL: NCT00707889
Title: An Open-Label, Randomized Phase 2 Study of ABT-869 in Combination With mFOLFOX6 (Oxaliplatin, 5-Fluorouracil, and Folinic Acid) Versus Bevacizumab in Combination With mFOLFOX6 as Second-line Treatment of Subjects With Advanced Colorectal Cancer
Brief Title: Phase 2 Study of ABT-869 in Combination With mFOLFOX6 Versus Bevacizumab in Combination With mFOLFOX6 to Treat Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-300; 2007-007081-38 (EudraCT Number); NCT00788411 (obsolete NCT alias)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Advanced Colorectal Cancer; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — linifanib; Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Open-label to Bevacizumab plus mFOLFOX6
  Interventions: Drug: bevacizumab; Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil
- B (Active Comparator): Open-label to High-dose ABT-869 arm plus mFOLFOX6
  Interventions: Drug: ABT-869; Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil
- C (Active Comparator): Open-label to low-dose ABT-869 arm plus mFOLFOX6
  Interventions: Drug: oxaliplatin; Drug: folinic acid; Drug: fluorouracil; Drug: ABT-869

INTERVENTIONS:
Drug: ABT-869 — 12.5 mg QD, tablets taken orally days 1-14 of every 14-day cycle
  Arms: B
Drug: bevacizumab — 10 mg/kg QD, IV on Day 1 of each 14-day cycle
  Arms: A
Drug: oxaliplatin — 85 mg/m2 IV, 120 minutes on Day 1 of each 14-day cycle
  Other Names: mFOLFOX6 regimen
Drug: folinic acid — 400 mg/m2 IV, 120 minutes on Day 1 of each 14-day cycle
  Other Names: mFOLFOX6 regimen
Drug: fluorouracil — 400 mg/m2 IV bolus on Day 1 of each 14-day cycle; followed by 2400 mg/m2 IV infusion 46-48 hours
  Other Names: mFOLFOX6 regimen
Drug: ABT-869 — 7.5 mg QD tablets taken orally days 1-14 of every 14-day cycle
  Arms: C

SUMMARY:
To determine the effect of ABT-869 plus mFOLFOX6 compared to bevacizumab plus mFOLFOX6 on disease progression in advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Subject must be >/= 18 years of age. Subject (male or female) must be diagnosed with adenocarcinoma of the colon or rectum. Subject must have metastatic disease or locally recurrent disease that is not amenable to surgical resection with curative intent.

Subject must have received one prior chemotherapy regimen containing irinotecan or a fluoropyrimidine for locally recurrent or metastatic colon or rectal cancer.

Subject has experienced progressive disease during or following the previous anti-tumor treatment.

Subject may have received prior adjuvant treatment for colorectal cancer. Subject has measurable disease by RECIST criteria (randomized portion only). Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1. Subject must have adequate bone marrow, renal and hepatic function. Subject must have Partial Thromboplastin Time (PTT) < 1.5 x Upper Limit of Normal (ULN) and International Normalized Ratio (INR) < 1.5.

Exclusion Criteria:

Subject has received more than one prior therapy in the metastatic setting. Lead-in Cohort only: The subject may have received more than one prior therapy in the metastatic setting.

Subject has received cytotoxic chemotherapy within 21 days prior to Study Day 1.

Subject has received non-cytotoxic, anti-cancer therapy within 21 days or within a period defined by 5 half lives whichever is shorter, prior to Study Day 1.

Subject has not recovered to less than or equal to Grade 1 clinically significant adverse effects/toxicities of the previous therapy.

Subject has received prior treatment with a tyrosine kinase inhibitor targeting VEGF or PDGF.

Subject has received prior treatment with oxaliplatin in the metastatic setting. Lead-in cohort only: Prior treatment with oxaliplatin will be allowed provided that any neuropathy as a result of the oxaliplatin treatment has resolved to less than or equal to Grade 1.

Subject has had major surgery within 28 days of Study Day 1. Subject has had radiotherapy within 14 days of Study Day 1. Subject has a history of hypersensitivity to recombinant murine monoclonal antibodies, oxaliplatin or other platinum-containing compounds, fluorouracil, or folinic acid.

Subject has a known intolerance to bevacizumab. Subject has untreated brain or meningeal metastases. Subject is receiving therapeutic anticoagulation therapy . Subject has a history of/or currently exhibits clinically significant cancer related events of bleeding.

Subject currently exhibits symptomatic or persistent, uncontrolled hypertension.

Subject has a history of myocardial infarction, stroke, or transient ischemic attack within six months of Study Day 1.

History of another active cancer within the past 5 years except cervical cancer in situ, in situ carcinoma of the bladder, squamous cell or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Radiographic evaluation every 2 months, clinial evaluation every 2 weeks

SECONDARY OUTCOMES:
Overall survival | from randomization until patient death or alive at 5 years
12-month overall survival rate | from randomization until patient death or alive at 5 years
Objective response rate | from randomization until patient death or alive at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. McKee, MD, Study Director — AbbVie
Locations (46):
- United States (3):
  - Site Reference ID/Investigator# 11341, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 20801, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 8360, Nashville, Tennessee
- Australia (2):
  - Site Reference ID/Investigator# 18581, Bedford Park
  - Site Reference ID/Investigator# 23443, Herston
- Belgium (4):
  - Site Reference ID/Investigator# 18023, Bonheiden
  - Site Reference ID/Investigator# 23646, Brussels
  - Site Reference ID/Investigator# 18026, Leuven
  - Site Reference ID/Investigator# 18022, Roeselare
- Brazil (2):
  - Site Reference ID/Investigator# 26662, Jaú
  - Site Reference ID/Investigator# 24245, Porto Alegre
- Canada (3):
  - Site Reference ID/Investigator# 23265, Barrie
  - Site Reference ID/Investigator# 21083, Edmonton
  - Site Reference ID/Investigator# 22465, Ottawa
- Site Reference ID/Investigator# 22141, Náchod, Czechia
- Greece (3):
  - Site Reference ID/Investigator# 22289, Heraklion
  - Site Reference ID/Investigator# 22286, Thessaloniki
  - Site Reference ID/Investigator# 22287, Thessaloniki
- Site Reference ID/Investigator# 20281, Wellington South, New Zealand
- Poland (3):
  - Site Reference ID/Investigator# 20141, Olsztyn
  - Site Reference ID/Investigator# 17946, Warsaw
  - Site Reference ID/Investigator# 38284, Warsaw
- Portugal (4):
  - Site Reference ID/Investigator# 23908, Aveiro
  - Site Reference ID/Investigator# 22324, Coimbra
  - Site Reference ID/Investigator# 23724, Faro
  - Site Reference ID/Investigator# 23964, Lisbon
- Romania (7):
  - Site Reference ID/Investigator# 23303, Baia Mare
  - Site Reference ID/Investigator# 23302, Brasov
  - Site Reference ID/Investigator# 17962, Bucharest
  - Site Reference ID/Investigator# 17964, Bucharest
  - Site Reference ID/Investigator# 23304, Bucharest
  - Site Reference ID/Investigator# 17961, Cluj-Napoca
  - Site Reference ID/Investigator# 23305, Craiova
- Russia (4):
  - Site Reference ID/Investigator# 24422, Moscow
  - Site Reference ID/Investigator# 25063, Moscow
  - Site Reference ID/Investigator# 25065, Moscow
  - Site Reference ID/Investigator# 24423, Moscow
- South Korea (3):
  - Site Reference ID/Investigator# 18281, Seoul
  - Site Reference ID/Investigator# 18283, Seoul
  - Site Reference ID/Investigator# 18282, Seoul
- Spain (6):
  - Site Reference ID/Investigator# 22809, A Coruña
  - Site Reference ID/Investigator# 22807, Barcelona
  - Site Reference ID/Investigator# 22804, Madrid
  - Site Reference ID/Investigator# 22801, Madrid
  - Site Reference ID/Investigator# 22803, Pamplona Navarra
  - Site Reference ID/Investigator# 22800, Santander